CLINICAL TRIAL: NCT03456401
Title: Activity and Safety of Third Line Tyrosin Kinase Inhibitor (TKI) After 2 Tyrosin Kinase Inhibitors (TKIs) in Patients With Metastatic Renal Cell Carcinoma (mRCC) (Tokio Study)
Brief Title: Third Line TKI After 2 TKIs in Patients With mRCC (Tokio Study)
Acronym: TOKIO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: availability of new and more promising therapeutic agents than expected in the experimentation in question
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001956-52
Record Dates: First submitted 2014-11-11; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Renal Cancer Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib or Sunitinib (Other): Sorafenib will be administered at 400 mg bid daily Sunitinib will be administered at 50 mg die orally (4 week on/2 weeks off)
  Interventions: Drug: Sorafenib or Sunitinib

INTERVENTIONS:
Drug: Sorafenib or Sunitinib — After two lines of TKIs, patients received a third line with sunitinib or sorafenib, according to previous treatments
  Other Names: Nexavar or Sutent

SUMMARY:
The study aims to evaluate the efficacy of a third TKI after two previous lines of therapy with TKIs, in terms of median progression free survival (mPFS), in patients affected by metastatic renal cancer cell.

Patients receiving the sequence Sunitinib- Axitinib, will receive Sorafenib.

Patients receiving the sequence Pazopanib-Sorafenib, will receive Sunitinib.

Sorafenib dosage 400mg orally, twice a day.

Sunitinib dosage 50 mg 4 weeks on followed by 2 weeks a rest.

The therapy will be continued until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Advanced RCC presents poor prognosis, because his pathogenesis is not clearly understood.

Additionally, the Von Hippel Lindau (VHL) gene is mutated in the majority of sporadic and familial clear cell renal cancer. The mechanism by which VHL mutation leads to RCC development and progression is postulate to be in part thought production of the protein VEGF (Vascular Endothelial Grow Factor).

VEGF over-expression may be pertinent in RCC via multiple mechanism in addition to angiogenesis, including effects on dendritic cells and inhibition of apoptosis through preservation of cyclin dependent kinase inhibitors.

VEGF expression could represented an independent prognostic factors for survival possibly linking expression of this protein with clinical outcome.

Sunitinib and pazopanib are the standard therapy as first line in mRCC. At sunitinib failure a second line with axitinib or everolimus or sorafenib should be considered to improve the clinical outcome of the disease. Up to now there is not a clear evidence of superiority in favour of an agent versus the others available.

At pazopanib failure no evidences are available to support physicians in the decision making in the everyday clinical practice.

Moreover no data are available in third line with a TKi after two previous lines of therapy with TKIs.

This study was designed to evaluate prospectively the efficacy of two different sequences of TKis in third line:

The first (group A) to evaluate the efficacy of sorafenib after two previous lines of TKIs with sunitinib followed by axitinib

The second (group B) to evaluate the efficacy of sunitinib after two previous lines of TKIs with pazopanib followed by sorafenib.

400 mg bid is the standard approved dose for sorafenib in the treatment of mRCC while 50 mg for 4 consecutive weeks every six weeks is the standard dose for sunitinb

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with histological diagnosis of Renal Cell Carcinoma (RCC)
* Measurable disease
* Previous treatment with two sequences of TKIs including sunitinib followed by axitinib and pazopanib followed by sorafenib.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0 or 1
* All prognostic group according to Heng criteria
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hemoglobin > or equal to 10.0 g/dl
  * Absolute neutrophil count (ANC) >1,500/mm3
  * Platelet count > or equal to 100,000/ml
  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * ALT (Alanine Transferase) and AST (Aspartate transferase) ≤ 2.5 x upper normal limit (ULN)
  * ALP (Alkaline phosphatase) ≤ 4 x ULN
  * PT-INR/PTT (Protrombine Time; International Normalized Ratio; Partial Tromboplastine Time)≤ 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.] For patients on warfarin, close monitoring of at least weekly evaluations will be performed, until INR is stable based on a measurement at pre-dose, as defined by the local standard of care.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Previous treatment for metastatic RCC other than pazopanib followed by sorafenib or sunitinib followed by axitinib
* History of cardiac disease: congestive heart failure >NYHA class 2 (New York Heart Association); active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension (>= 160 mmHg systolic and/or 90 mmHg diastolic).
* History of HIV infection
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dyalisis
* History of other disease, metabolic dysfunction, physical examination findings or clinical laboratory findings giving reasonable suspicion of a disease condition that contraindicates use of an investigational drug or patient at high risk from treatment complications
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 2 years prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
median progression free survival (mPFS) | up to five years
  To evaluate the efficacy of a third TKI after two previous lines of therapy with TKIs, in terms of mPFS; time from the first treatment administration to first disease progression or death (months). It will be evaluated up to five years.

SECONDARY OUTCOMES:
OS (Overall Survival) | up to five years
  To evaluate overall survival: time from first treatment to death (months) (up to five years).
safety of a third line TKI | up to five years
  To evaluate the safety of a third line TKI; it will be evaluated and graded according to NCI-CTC version 3.0 criteria (Common Toxicity Criteria). Adverse events will be registered since treatment starts until end of treatment visit (30 +/- 7 days after end of treatment)
Quality of life through specific questionnaire EORTC QLQ-C30 | up to five years
Quality of life through specific questionnaire FKSI-19 | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Study Chair — IRCCS Istituto Nazionale Tumori
Locations (1):
- Istituto Tumori, Milan, Mi, Italy